CLINICAL TRIAL: NCT04881643
Title: Facilitating Implementation of Evidence-based Psychological Therapy for Posttraumatic Stress Disorder in Health Care Services Through a Digital Support - A Feasibility Study
Brief Title: Blended Treatment för PTSD Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Sigrid Salomonsson, Principal Investigator and PhD, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: dnr P2020/46
Record Dates: First submitted 2021-05-03; First posted 2021-05-11 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Acceptability of Health Care
Keywords: cbt; PTSD; digital support
MeSH Terms: conditions — Patient Acceptance of Health Care; Color Vision Defects; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Feasibility and pilot study using within-group design. 20 patients will be included and 4 therapists. Semi-structured interviews will be conducted after treatment with a selection of therapists and patients with questions regarding the helpfulness and feasibility of the treatment. Effects of treatment patients estimate forms regarding PTSD, depression, anxiety, sleep, quality of life, function and patient satisfaction / acceptance. Measurements are performed before, during, immediately after and 6 months after treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blended treatment for PTSD (Experimental): A trauma-focused CBT where internet-based treatment is blended with face-to-face sessions with a therapist.
  Interventions: Behavioral: Trauma-focused cognitive behavioural therapy via a digital support

INTERVENTIONS:
Behavioral: Trauma-focused cognitive behavioural therapy via a digital support — A blended treatment approach to PTSD, blending internet-based CBT with face-to-face sessions with a therapist

SUMMARY:
Feasibility and pilot study using within-group design with the aim of examining whether the blended psychological treatment for PTSD is acceptable for patients and therapists. 20 patients will be included and 4 therapists. Semi-structured interviews will be conducted after treatment with a selection of therapists and patients with questions regarding the helpfulness and feasibility of the treatment. Effects of the treatment will be assessed via standardized self-report outcome measures regarding PTSD, depression, anxiety, sleep, quality of life, function and patient satisfaction / acceptance. Measurements are conducted before, during, immediately after and 6 months after treatment. The study is conducted at 2 psychiatric outpatient clinics in the Stockholm Region.

DETAILED DESCRIPTION:
Research question and hypothesis

The research question is: Is blended psychological treatment for PTSD via a digital support acceptable and applicable to patients and clinicians? The hypothesis is that testing the digital support and blended delivery format in a smaller scale pilot study will bring to light how the support and treatment could be augmented to better adhere to patients and clinicians needs.

Procedure

The feasibility study will be carried out in collaboration with 2 psychiatric care units in the Stockholm region. In these clinics a handful of therapists will implement the treatment with altogether 20 PTSD patients and assess the digital support and treatment modules. A task group of 3 psychologists will develop the treatment platform and the inherent modules and work materials. The therapists will work closely with the task group and regularly provide feedback of their experiences of working with the platform. Learning obtained from the study will be utilized to improve and adjust the digital support and treatment procedure in preparation for a larger randomized study.

To enable implementation of the digital support in health care services it will be integrated into the digital health care platform Support and Treatment (SOB). SOB is a well-established national health system available to clinicians via the patient medical journals. The support will be internet-based and consist of self-help modules that incorporates similar treatment components as those found in evidence-based trauma-focused cognitive behavioural therapy (TF-CBT) protocols. The treatment modules will consist of educational texts, filmed illustrations, case examples, and relevant worksheets. The purpose of the support is to function as a treatment foundation, both for face-to-face appointments and as guided self-help.

Methodology/approach/data analysis

To be included in the study participants must meet diagnostic criteria for PTSD as their primary problem according to Diagnostic and Statistical Manual of Mental Disorders (DSM-5), have basic reading and writing skills in Swedish, and not express acute suicidal ideation. Patients with concurrent comorbid psychiatric problems are eligible for inclusion unless another psychiatric diagnosis is assessed as primary to PTSD. Patients will be recruited from the regular flow of patients who seek treatment for psychological problems in the selected clinics.

The research question will be investigated using both qualitative and quantitative research methods. Qualitative data will be collected via semi-structured interviews with therapists and a selection of patients with the aim of exploring participant's experience of working with the program and strengths and weaknesses of the blended treatment package. Interviews will be carried out by members of the research group post-treatment. The interviews will be transcribed and thematically analyzed.

To further assess patient acceptability two questionnaires will be distributed following treatment. The Client Satisfaction Questionnaire-8 (CSQ-8) has demonstrated good psychometric properties including high reliability and construct validity. The Credibility/Expectancy Questionnaire (CEQ) is the most widely used measure of treatment credibility and expectancy in psychotherapy research. The CEQ consists of five items that are scored on a 10-point likert scale and has demonstrated high internal consistency (Cronbach's α = .84) and high test-retest reliability (r = .75 - .83). Treatment effects in terms of PTSD-symptoms, other psychiatric symptoms, general functioning and quality of life, will be measured by standardized self-rated measures with good reliability and validity. Outcome measures will be administered before, during and after therapy. Statistical analysis will be conducted to measure change over time and effect sizes (hedges g) will be calculated. Moreover, reliable change (RC) and clinically significant change (CSC) will be meassured according to the criteria established by Jacobson and Truax (22).

Significance

The purpose of this project is to increase availability to evidence-based treatment for individuals with PTSD that is effective, acceptable and resource-efficient. PTSD patients make up 2.8% (n = 10342) of the total number of psychiatric patients in the Stockholm region in 2018, according to data collected via the project "dissemination of guideline based care for PTSD". Of these, 15-20% of patients are estimated to have received evidence-based psychological treatment. This indicates that the majority of individuals suffering from PTSD are not receiving appropriate care in Stockholm. Blended treatment may be a solution to this problem and that a small scale feasibility/pilot study is a valuable first step to test the treatment and learn how it can be improved before launching a larger randomized trial. Hence the significance of this study.

ELIGIBILITY:
Inclusion Criteria:

* PTSD according to DSM-5 criteria (American Psychiatric Association, 2013) as a primary problem
* have basic knowledge of speaking and writing in Swedish,
* not undergo other psychological treatment for PTSD during the course of the study;
* be at least 18 years old
* not be exposed to ongoing violence or threats
* if antidepressants for depression / anxiety are available, the dose must have been stable for at least 6 weeks before starting treatment.

Patients who express an interest in participating receive information about the study. Patients who subsequently carry out the assessment and meet the inclusion criteria receive accurate oral and written information about what participation includes and handling of personal data and data. If the patient wants to participate and gives written consent, the person is included in the study.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-12-04 (Actual); Study Completion 2023-07-03 (Actual)

PRIMARY OUTCOMES:
Acceptability of treatment among patients and therapists | Post treatment, 12-20 weeks after enrollment
  Semi-structured interviews

SECONDARY OUTCOMES:
The Client Satisfaction Questionnaire-8 (CSQ-8) | post treatment, 8-12 weeks after enrollment
  Self rated satisfaction of treatment. Minimum value 8, maximum value 32 where higher values indicate greater satisfaction with the treatment.
The Credibility/Expectancy Questionnaire (CEQ) | Week 1 of treatment
  Self rated Credibility of treatment. Minimum value 3, maximum value 27 for each factor, where higher values indicate greater Credibility/Expectancy of the treatment.
The Posttraumatic stress disorder checklist 5 (PCL-5) | Pre-treatment, weekly, post treatment 8-12 weeks after enrollment, and 6-month follow up
  Self rated PTSD-symptoms. Minimum value 0, maximum value 80, where higher values indicate more PTSD symptoms.
Patient Health Questionnaire 9 (PHQ-9) | Pre-treatment, weekly, post treatment 8-12 weeks after enrollment, and 6-month follow up
  Self rated depressive symptoms. Minimum value 0, maximum value 27, where higher values indicate more depressive symptoms.
Generalised Anxiety Disorder 7-item scale (GAD-7) | Pre-treatment, Post treatment 8-12 weeks after enrollment, and 6-month follow up
  Self rated anxiety symptoms. Minimum value 0, maximum value 21, where higher values indicate more anxiety symptoms.
Insomnia Severity Index (ISI) | Pre-treatment, Post treatment 8-12 weeks after enrollment, and 6-month follow up
  Self rated insomnia symptoms. Minimum value 0, maximum value 28, where higher values indicate more insomnia symptoms.
Brunnsviken Brief Quality of Life Questionnaire (BBQ) | Pre-treatment, Post treatment 8-12 weeks after enrollment, and 6-month follow up
  Self rated quality of life. Minimum value 0, maximum value 96, where higher values indicate higher quality of life satisfaction.
World health organization disability assessment schedule (WHODAS 2.0) | Pre-treatment, Post treatment 8-12 weeks after enrollment, and 6-month follow up
  Self rated disability. Minimum value 0, maximum value 100, where higher values indicate more disability.
Negative effects questionnaire (NEQ 20) | Post treatment 8-12 weeks after enrollment
  Self rated negative effects of treatment. Minimum value 0, maximum value 80, where higher values indicate more negative effects.
Internet Intervention Patient Adherence Scale (IIPAS) | Post treatment 8-12 weeks after enrollment
  Therapist-rated questionnaire regarding patient adherence to an internet-delivered psychological treatment. The scale consists of 5 items rated from 0-4 with higher ratings indicating greater adherence. Total range of scale is 0-20.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lundin J, Jansson-Frojmark M, Gustafsson-Bjorverud L, Grey N, Santoft F, Ehlers A, Carlbring P, Lundgren T, Bragesjo M, Salomonsson S. Integrating digital and in-person therapy for PTSD: feasibility and acceptability of blended trauma-focused cognitive therapy in routine care. Front Psychiatry. 2024 Sep 5;15:1447651. doi: 10.3389/fpsyt.2024.1447651. eCollection 2024. PMID 39301223